CLINICAL TRIAL: NCT01034280
Title: Epidemiological Study of Trisomy 21 With Research of Correlations Between Phenotype (Physical, Psychometrical) and Genotype (Genome, Transcriptome, Proteome)
Brief Title: Correlations Phenotype / Genotype in Down Syndrome
Acronym: INTREPID
Status: Completed | Type: Observational
Sponsor: Institut Jerome Lejeune (Other)
Collaborators: Fondation Jérôme Lejeune (Other)
Responsible Party: Sponsor
Other Study IDs: IJL-PG-EP03; Intrepid
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2009-12

CONDITIONS: Down Syndrome
Keywords: Down Syndrome; phenotype; genotype; patient family
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
The purpose of this study is to correlate phenotype and genotype of Down syndrome patients in order to identify the biochemical reactions involved in their mental retardation and their other phenotypic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Down syndrome patients
* age: 8years and older
* assessment by the psychometric tests
* possible blood tests

Exclusion Criteria:

* no exclusion criteria

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Down syndrome patients
Sampling Method: Probability Sample
Enrollment: 524 (Actual)
Dates: Start 2004-03; Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yann Grattau, M.D., Study Director — Institut Jerome Lejeune
Locations (1):
- Institut Jerome Lejeune, Paris, France